CLINICAL TRIAL: NCT04020185
Title: Phase I/IIA Safety and Efficacy Study of IMSA101 in Patients With Advanced Treatment-Refractory Malignancies
Brief Title: Safety and Efficacy Study of IMSA101 in Refractory Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ImmuneSensor Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMSA101-101
Record Dates: First submitted 2019-07-11; First posted 2019-07-15 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — Immune Checkpoint Inhibitors; Jupiter; Therapeutics

STUDY DESIGN:
Intervention Model Description: Phase I includes a monotherapy arm and an immune checkpoint inhibitor (ICI) combination therapy arm Phase II includes three arms, Arm A monotherapy, Arm B immuno-oncology (IO) combination therapy, Arm C IO combination therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Ph I Monotherapy (Experimental): * Dose escalation design in which administered dose levels of IMSA101 as monotherapy will be escalated stepwise in successive cohorts of 3 to 6 patients per dose group (using a standard 3+3 study design) of IMSA101 until the RP2D or maximum tolerated dose (MTD) level is identified.
  * The first patient enrolled in each dose level must complete the first two weeks of Cycle 1 prior to enrolling the second and third patients.
  * Dose levels to be evaluated include (although not necessarily limited to) 100 µg (representing 1/60th of the pre-clinical Highest Non-Severely Toxic Dose [HNSTD] dose), 200 µg, 400 µg, 800 µg, and 1,200 µg.
  Interventions: Drug: IMSA101
- Ph I Combination Therapy (Experimental): * Ph I combination dosing of IMSA101 shall be evaluated upon satisfaction of the following criteria:
    * A given dose level (combo dose level 1) has been confirmed as safe for monotherapy dosing (i.e. 2/6 patients experience Cycle 1 DLT).
    * The next higher dose level (combo dose level 2) has been confirmed as safe for monotherapy dosing (i.e. 2/6 patients experience Cycle 1 DLT).
    * The dose level (combo dose level 1) is found to demonstrate adequate IMSA101 pharmacodynamic (PD) activity based on exploratory endpoints.
  * Eligible patients shall have demonstrated RECIST stable disease through ≥ 4 consecutive cycles of an approved PD-1/PD-L1-targeted ICI with no Grade ≥ 3 CTCAE events considered to be drug-related.
  * Safety evaluations and dose escalation of IMSA101 administered in combination with current therapy shall proceed in a manner consistent with monotherapy escalation and shall proceed independently of monotherapy dose escalation.
  Interventions: Drug: IMSA101; Drug: Immune checkpoint inhibitor (ICI)
- Ph II Monotherapy (Arm A) (Experimental): * This dose-expansion arm of 20 patients is intended to confirm the tolerability of the RP2D and identify provocative signals of IMSA101 anti-tumor activity when administered as monotherapy
  * Tumor type to be evaluated will be identified prior to Phase IIA commencement and will be documented in a protocol amendment.
  Interventions: Drug: IMSA101
- Ph II Combination Therapy (Arm B) (Experimental): * This dose-expansion arm of 20 patients is intended to confirm the tolerability of the RP2D and identify provocative signals of IMSA101 anti-tumor activity when administered as combination therapy with PD-1/PD-L1 targeted immune checkpoint inhibitors.
  * This arm shall include a safety run-in of 5-10 patients.
  * Tumor type and corresponding treatment combination will be identified prior to Phase IIA commencement and documented in a protocol amendment.
  Interventions: Drug: IMSA101; Drug: Immune checkpoint inhibitor (ICI)
- Ph II Combination Therapy (Arm C) (Experimental): * This dose-expansion arm of 20 patients is intended to confirm the tolerability of the RP2D and identify provocative signals of IMSA101 anti-tumor activity when administered as combination therapy with non-PD-1/PD-L1-targeted immuno-oncology (IO) drugs approved by the FDA.
  * This arm shall include a safety run-in of 5-10 patients.
  * Tumor type and corresponding treatment combination will be identified prior to Phase IIA commencement and documented in a protocol amendment..
  Interventions: Drug: IMSA101; Drug: Immuno-oncology (IO) therapy

INTERVENTIONS:
Drug: IMSA101 — IMSA101 administered by intra-tumoral (IT) injection on Day 1 of Weeks 1, 2, and 3 for Cycle 1 and on Day 1 of Weeks 1 and 3 for all subsequent cycles.
Drug: Immune checkpoint inhibitor (ICI) — Administered according to product label
  Arms: Ph I Combination Therapy; Ph II Combination Therapy (Arm B)
Drug: Immuno-oncology (IO) therapy — Administered according to product label
  Arms: Ph II Combination Therapy (Arm C)

SUMMARY:
Open-label, dose escalation (Phase I) and dose expansion (Phase IIA) study of patients receiving intra-tumoral IMSA101 alone or in combination with an immune checkpoint inhibitor (ICI) (Phase I and II)

DETAILED DESCRIPTION:
This is an open-label, dose escalation (Phase I), and dose expansion (Phase IIA) study designed to evaluate safety and efficacy of IMSA101 alone or in combination with an ICI (Phase I and II). Therefore, the study will be conducted in 2 phases. The dose of IMSA101 in Phase IIA will be based on the monotherapy and combination Recommended Phase 2 Doses (RP2Ds) from Phase I.

The following methodology applies to all patients (unless otherwise indicated):

* Pre-treatment screening radiographic tumor assessments will be collected within 30 days prior to initial dose for all patients. Photographic assessments for cutaneously-accessible lesions will be performed as detailed in a separate photography manual.
* Treatment cycles will be 28 days in duration with lesions injected weekly on Day 1 for the first three weeks of Cycle 1 and then every 2 weeks during cycles 2 and beyond.
* A single pre-defined lesion/lesion site (longest diameter ≥ 10 mm and ≤ 35 mm) shall be injected throughout study duration, if possible. Where the original injection site is considered by the investigator to become inaccessible, a second lesion/lesion site shall be selected as a replacement and this shall be used henceforth so long as it is considered accessible. Subsequent injection sites shall be replaced when they are considered inaccessible.
* Where no remaining accessible lesions are present and where benefit of IMSA101 therapy is, in the opinion of the investigator, being derived by the patient, continued injections of IMSA101 into the vicinity of an inaccessible lesion or, in the case that a lesion can no longer be radiographically visualized, into the last known location of the non-visible lesion shall be allowed.
* Patients will be admitted to the hospital for observation overnight following IT injection with IMSA101 on Day 1 of Cycle 1. Patients will be followed throughout the study for drug tolerability and safety by collection of clinical and laboratory data, including information on adverse events (AEs) using CTCAE v5.0 criteria, serious adverse events (SAEs), DLTs, concomitant medications, vital signs, and electrocardiograms (ECGs).
* Patients will be assessed for anti-tumor efficacy based on radiographic assessments and if applicable, photographic tumor assessments, and analysis of Objective Response Rate (ORR), Time to Progression (TTP), and Progression Free Survival (PFS) using RECIST criteria (Appendix 13.2) at screening and the end (≤ 7 days) of even numbered cycles (Cycle 2, Cycle 4, etc.) after the first dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent and mental capability to understand the informed consent
2. Male or female patients > 18 years of age
3. Histologically or cytologically documented locally advanced or metastatic solid tumor malignancies refractory to or otherwise ineligible for treatment with standard-of-care agents/regimens, including but not limited to:

   * Malignant melanoma
   * Hormone receptor negative breast cancer
   * Gastro-esophageal cancer
   * Non-small cell lung cancer
   * Head and neck cancer
   * Hepatoma
   * Renal cell carcinoma
4. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1
5. Evaluable or measurable disease as follows:

   * A minimum of 3 RECIST-evaluable lesions: one that is suitable for injection and biopsied; one non-injected that will be biopsied for abscopal effect; and one measurable lesion that will be followed for response only.
   * Injectable tumors shall be accessed by intralesional (cutaneous) or percutaneous injection only, including those lesions that are visible, palpable, or detectable by standard radiographic or ultrasound methods. Neither surgical procedures nor endoscopically-guided injections including those to endobronchial, endoluminal, or endosinusial spaces shall be allowed. While no anatomic locations are required or disallowed, lesions selected for intratumoral injection must, in the opinion of the investigator:
   * Not be immediately adjacent to blood vasculature or other physiologic landmarks in such a way that will accrue undue safety risk to the patient
   * Have longest diameter ≥ 10 mm and ≤ 50 mm
   * Be fully efficacy evaluable per RECIST v1.1 criteria
6. Life expectancy > 3 months (Phase I) and > 6 months (Phase IIA)
7. ECG without evidence of clinically meaningful conduction abnormalities or active ischemia as determined by the investigator
8. Acceptable organ and marrow function as defined below:

   * Absolute neutrophil count > 1,500 cells/μL
   * Platelets > 50,000 cells/μL
   * Total bilirubin ≤ 1.5 times the upper limit of normal (ULN)
   * Aspartate aminotransferase (AST)/alanine transaminase (ALT) ≤ 2.5 times ULN. If liver metastases are present, AST/ALT < 5 times ULN
   * Serum creatinine < 1.5 mg/dL and a measured creatinine clearance ≥ 50 mL/min using the Cockcroft-Gault formula
   * Prothrombin time (PT)/partial thromboplastin time (PTT) ≤ 1.5 times ULN
9. Women of child-bearing potential (defined as a female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or is not postmenopausal (defined as amenorrhea for at least 12 consecutive months with an appropriate clinical profile at the appropriate age, e.g., greater than 45 years) must have a negative serum pregnancy test prior to first dose of study drug
10. Male and female patients with reproductive potential must agree to use two forms of highly effective contraception throughout the study
11. Phase I combination only: Demonstrated RECIST stable disease through ≥ 4 consecutive cycles of an approved PD-1 or PD-L1 targeted ICI with no Grade ≥ 3 CTCAE events considered by the investigator to be drug-related.

Exclusion Criteria:

1. Anti-cancer therapy within 4 weeks or < 5 half-lives of the first dose of study drug.
2. Failure to recover to Grade 1 or less from clinically significant AEs due to prior anti-cancer therapy.
3. Known untreated brain metastases or treated brain metastases that have not been stable (scan showing no worsening of central nervous system (CNS) lesion[s] and no requirement of corticosteroids) ≥ 4 weeks prior to study enrollment
4. Baseline prolongation of QT/QTc interval (QTc interval > 470)
5. Uncontrolled intercurrent illness (including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations) that in opinion of the investigator would limit compliance with study requirements
6. Women who are pregnant or breastfeeding
7. Phase I combination only: Prior tumor progression through PD-1 or PD-L1 targeted ICI therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa S Mooneyham, Study Director — Vice President, ImmuneSensor Therapeutics Inc.
Locations (6):
- United States (6):
  - Honor Health, Scottsdale, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Northwestern University, Chicago, Illinois
  - Atlantic Health System/Morristown Medical Center, Morristown, New Jersey
  - UT Southwestern, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jacoby J, Mahalingam D, Alistar A, Garmey E, Kazmi S, Mooneyham T, Sun L, Yap TA, Vu P, Moser J. Phase 1 first-in-human dose-escalation study of IMSA101, a novel cyclic di-nucleotide STING agonist, for patients with advanced solid tumor malignancies. J Immunother Cancer. 2025 Jun 18;13(6):e011572. doi: 10.1136/jitc-2025-011572. PMID 40533265

RESULTS

PARTICIPANT FLOW:
Groups:
- Monotherapy 100 μg: 100 μg of IMSA101 injected intra-tumorally weekly on Day 1 for the first 3 week cycles of Cycle 1, and then every 2 weeks during Cycles 2 and beyond.
- Monotherapy 200 μg: 200 μg of IMSA101 injected intra-tumorally weekly on Day 1 for the first 3 week cycles of Cycle 1, and then every 2 weeks during Cycles 2 and beyond.
- Monotherapy 400 μg: 400 μg of IMSA101 injected intra-tumorally weekly on Day 1 for the first 3 week cycles of Cycle 1, and then every 2 weeks during Cycles 2 and beyond.
- Monotherapy 800 μg: 800 μg of IMSA101 injected intra-tumorally weekly on Day 1 for the first 3 week cycles of Cycle 1, and then every 2 weeks during Cycles 2 and beyond.
- Monotherapy 1200 μg: 1200 μg of IMSA101 injected intra-tumorally weekly on Day 1 for the first 3 week cycles of Cycle 1, and then every 2 weeks during Cycles 2 and beyond.
- Combination Therapy 800 μg: 800 μg of IMSA101 injected intra-tumorally weekly on Day 1 for the first 3 week cycles of Cycle 1, and then every 2 weeks during Cycles 2 and beyond.
  Plus an approved ICI administered as per product label.
- Combination Therapy 1200 μg: 1200 μg of IMSA101 injected intra-tumorally weekly on Day 1 for the first 3 week cycles of Cycle 1, and then every 2 weeks during Cycles 2 and beyond.
  Plus an approved ICI administered as per product label.
- Combination Therapy 2400 μg: 2400 μg of IMSA101 injected intra-tumorally weekly on Day 1 for the first 3 week cycles of Cycle 1, and then every 2 weeks during Cycles 2 and beyond.
  Plus an approved ICI administered as per product label.
Period: Overall Study
Arm/Group | Monotherapy 100 μg | Monotherapy 200 μg | Monotherapy 400 μg | Monotherapy 800 μg | Monotherapy 1200 μg | Combination Therapy 800 μg | Combination Therapy 1200 μg | Combination Therapy 2400 μg
Started | 4 | 3 | 4 | 4 | 7 | 4 | 7 | 7
Completed | 3 | 2 | 3 | 2 | 4 | 4 | 4 | 5
Not Completed | 1 | 1 | 1 | 2 | 3 | 0 | 3 | 2
Not completed — Death | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0
Not completed — Consent withdrawn | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Not completed — Patient in hospice | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Continuing on expanded access | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Patients who received at least 1 dose of IMSA101.
Groups:
- Combination Therapy 800 μg: 800 μg of IMSA101 injected intra-tumorally weekly on Day 1 for the first 3 week cycles of Cycle 1, and then every 2 weeks during Cycles 2 and beyond.
  Plus an ICI administered as per product label.
- Combination Therapy 1200 μg: 1200 μg of IMSA101 injected intra-tumorally weekly on Day 1 for the first 3 week cycles of Cycle 1, and then every 2 weeks during Cycles 2 and beyond.
  Plus an ICI administered as per product label.
- Combination Therapy 2400 μg: 2400 μg of IMSA101 injected intra-tumorally weekly on Day 1 for the first 3 week cycles of Cycle 1, and then every 2 weeks during Cycles 2 and beyond.
  Plus an ICI administered as per product label.
- Total: Total of all reporting groups
Arm/Group | Monotherapy 100 μg | Monotherapy 200 μg | Monotherapy 400 μg | Monotherapy 800 μg | Monotherapy 1200 μg | Combination Therapy 800 μg | Combination Therapy 1200 μg | Combination Therapy 2400 μg | Total
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 7 | 4 | 7 | 7 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 1 | 1 | 3 | 1 | 7 | 3 | 22
  >=65 years | 1 | 0 | 3 | 3 | 4 | 3 | 0 | 4 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (12.01) | 53.7 (2.08) | 66.5 (4.12) | 64.8 (6.95) | 65.0 (14.29) | 74.0 (11.34) | 50.3 (10.89) | 63.0 (21.53) | 61.4 (14.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 3 | 2 | 5 | 2 | 3 | 6 | 22
  Male | 3 | 3 | 1 | 2 | 2 | 2 | 4 | 1 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 2 | 7
  Not Hispanic or Latino | 3 | 2 | 3 | 3 | 7 | 3 | 4 | 5 | 30
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
  White | 3 | 1 | 1 | 2 | 5 | 4 | 4 | 6 | 26
  More than one race | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Unknown or Not Reported | 1 | 1 | 2 | 1 | 0 | 0 | 2 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities
Description: Highest dose level of IMSA101 at which no more than 1 out of 6 patients experienced a dose limiting toxicity (DLT) during the first cycle (28 days) of therapy.
Time Frame: Cycle 1 (28 days) of therapy
Population: Number of patients who received at least 3 doses of IMSA101 in Cycle 1 and completed 4 weeks on study, or received at least 1 dose of IMSA101 and experienced a DLT during Cycle 1 per dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Monotherapy 100 μg | Monotherapy 200 μg | Monotherapy 400 μg | Monotherapy 800 μg | Monotherapy 1200 μg | Combination Therapy 800 μg | Combination Therapy 1200 μg | Combination Therapy 2400 μg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 3 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Statistical Analysis 1: Comparison: Monotherapy 100 μg vs Monotherapy 200 μg vs Monotherapy 400 μg vs Monotherapy 800 μg vs Monotherapy 1200 μg vs Combination Therapy 800 μg vs Combination Therapy 1200 μg vs Combination Therapy 2400 μg; Test type: Other; maximum tolerated dose (monotherapy) = 1200

2. Secondary Outcome: Best Overall Response
Description: The sum of number of patients with best overall response (complete response, partial response, stable disease or progressive disease) as per RECIST v1.1 until End of Treatment. Tumor response was evaluated at the end of each even numbered cycle (eg. Cycle 2, Cycle 4, etc.) until End of Treatment.
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Monotherapy 100 μg | Monotherapy 200 μg | Monotherapy 400 μg | Monotherapy 800 μg | Monotherapy 1200 μg | Combination Therapy 800 μg | Combination Therapy 1200 μg | Combination Therapy 2400 μg
Number analyzed (Participants) | 4 | 3 | 3 | 2 | 6 | 4 | 5 | 4
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Stable Disease | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
  Progressive Disease | 4 | 3 | 2 | 2 | 6 | 3 | 4 | 3
  Not Evaluable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 9 months
Description: AE reporting began at the time of study treatment administration and continued until up to 30 days after the last dose, and ranged from to 28 to 261 days.
Groups:
- Monotherapy 800: 800 μg of IMSA101 injected intra-tumorally weekly on Day 1 for the first 3 week cycles of Cycle 1, and then every 2 weeks during Cycles 2 and beyond.
- Monotherapy 1200: 1200 μg of IMSA101 injected intra-tumorally weekly on Day 1 for the first 3 week cycles of Cycle 1, and then every 2 weeks during Cycles 2 and beyond.
- Combination Therapy 800 μg: 800 μg of IMSA101 injected intra-tumorally weekly on Day 1 for the first 3 week cycles of Cycle 1, and then every 2 weeks during Cycles 2 and beyond.
  Plus an ICI administered per product label.
- Combination Therapy 1200 μg: 1200 μg of IMSA101 injected intra-tumorally weekly on Day 1 for the first 3 week cycles of Cycle 1, and then every 2 weeks during Cycles 2 and beyond.
  Plus an ICI administered per product label.
- Combination Therapy 24000 μg: 2400 μg of IMSA101 injected intra-tumorally weekly on Day 1 for the first 3 week cycles of Cycle 1, and then every 2 weeks during Cycles 2 and beyond.
  Plus an ICI administered per product label.
Arm/Group | Monotherapy 100 μg | Monotherapy 200 μg | Monotherapy 400 μg | Monotherapy 800 | Monotherapy 1200 | Combination Therapy 800 μg | Combination Therapy 1200 μg | Combination Therapy 24000 μg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 1/4 | 2/4 | 1/7 | 0/4 | 1/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 2/4 | 1/3 | 2/4 | 3/4 | 1/7 | 1/4 | 5/7 | 5/7
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 4/4 | 3/4 | 7/7 | 4/4 | 7/7 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy 100 μg (N=4) | Monotherapy 200 μg (N=3) | Monotherapy 400 μg (N=4) | Monotherapy 800 (N=4) | Monotherapy 1200 (N=7) | Combination Therapy 800 μg (N=4) | Combination Therapy 1200 μg (N=7) | Combination Therapy 24000 μg (N=7)
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant bowel obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metastases to the CNS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy 100 μg (N=4) | Monotherapy 200 μg (N=3) | Monotherapy 400 μg (N=4) | Monotherapy 800 (N=4) | Monotherapy 1200 (N=7) | Combination Therapy 800 μg (N=4) | Combination Therapy 1200 μg (N=7) | Combination Therapy 24000 μg (N=7)
Injection site pain (General disorders) | 1 | 1 | 1 | 0 | 5 | 3 | 1 | 0
Fatigue (General disorders) | 1 | 3 | 3 | 1 | 3 | 1 | 3 | 5
Injection site erythema (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 1
Injection site dryness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site irritation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Odema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 4
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 3 | 1 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 3
Asthenia (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 3
Disease progression (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Injection site discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Performance status decreased (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Catheter site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 3 | 2
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 5 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Faeces discolored (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant bowel obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 1 | 1 | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 1 | 1 | 3 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 3 | 3
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemic seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Phantom pain (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to CNS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Shock (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/85/NCT04020185/Prot_SAP_000.pdf